CLINICAL TRIAL: NCT05858736
Title: Safety, Pharmacokinetics (PK) and Efficacy of AI-061, A 1:1 Co-formulation of AI-025 (Anti-PD-1) and ONC-392 (Anti-CTLA-4) Antibodies in Advanced Solid Tumors: An Open-Label Phase 1 Study
Brief Title: Safety, PK and Efficacy of AI-061 in Advanced Solid Tumors
Acronym: PRESERVE-009
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OncoC4, Inc. (Industry)
Collaborators: OncoC4 AU Pty Ltd (Unknown); Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AI-061-AU-01
Record Dates: First submitted 2023-05-03; First posted 2023-05-15 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Melanoma; Non Small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma; High Grade Serous Adenocarcinoma of Ovary; Primary Peritoneal Carcinoma; Fallopian Tube Cancer; Endometrial Cancer; Cervical Cancer; Renal Cell Carcinoma; Bladder Cancer; Esophageal Cancer; Gastric Cancer; Gastroesophageal-junction Cancer; Colorectal Cancer; Anal Cancer; Hepatocellular Carcinoma; Bile Duct Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Fallopian Tube Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Renal Cell; Urinary Bladder Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Colorectal Neoplasms; Anus Neoplasms; Carcinoma, Hepatocellular; Bile Duct Neoplasms

STUDY DESIGN:
Intervention Model Description: Three dose levels will be tested sequentially.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Level 1 (Experimental): AI-061, 200 mg, intravenous infusion, Q3W, up to 17 cycles or approximately 1 year.
  Interventions: Drug: AI-061
- Level 2 (Experimental): AI-061, 400 mg, intravenous infusion, Q3W, up to 17 cycles or approximately 1 year.
  Interventions: Drug: AI-061
- Level 3 (Experimental): AI-061, 600 mg, intravenous infusion, Q3W, up to 17 cycles or approximately 1 year.
  Interventions: Drug: AI-061

INTERVENTIONS:
Drug: AI-061 — A 1:1 Co-formulation of AI-025 (Anti-PD-1) and ONC- 392 (Anti-CTLA-4) Antibodies.
  Other Names: Anti-PD-1 and anti-CTLA-4 in 1:1 co-formulation

SUMMARY:
AI-061 is a co-formulation drug product (DP) consisting of 1:1 ratio mix of AI-025, an anti-PD-1 antibody, and ONC-392, an anti-CTLA-4 antibody. This is a dose escalation study to identify the maximum toxicity dose (MTD) or the recommended phase 2 dose (RP2D).

DETAILED DESCRIPTION:
AI-061 is a co-formulation drug product (DP) consisting of 1:1 ratio mix of AI-025, an anti-PD-1 antibody, and ONC-392, an anti-CTLA-4 antibody. Both CTLA-4 and PD-1 are known targets for immunotherapy. This Phase I study will test 3 fixed doses of AI-061 given as intravenous (IV) infusion, once every 21 days (q3w): 200 mg (consists of 100 mg ONC-392 and 100 mg AI-025), 400 mg and 600 mg. The target population is patient with advanced or metastatic solid tumors that progressed on standard care systemic therapy or intolerable to standard of care systemic therapy. The primary objective is to determine the maximum toxicity dose (MTD) or the Recommended Phase 2 dose (RP2D). The study design follows the classical 3+3 design for Phase 1 study that will enroll up to 18 subjects. The treatment will be terminated when patient has intolerable toxicity, or death, or disease progression, or complete of 17 cycles of treatment in approximate 1 year, whichever come first.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is greater or 18 years of age on the day of signing the informed consent.
2. All genders. Female subject with pregnancy potential must have a negative pregnancy test.
3. Patient must have a performance status of less than or equal to 1 on the ECOG Performance Scale.
4. Patients must have a histological or cytological diagnosis of solid tumors and have progressive locally advanced or metastatic disease.
5. Measurable disease as determined by RECIST v1.1 (either tumor lesion or lymph node lesion or both): Tumor mass: Must be accurately measurable in at least 1 dimension (longest diameter to be recorded) with a minimum size of: 10 mm by computed tomography (CT) scan (CT scan slide thickness must be less than 5 mm). Or: 20 mm by chest X-ray (if clearly defined and surrounded by aerated lung).

   Malignant lymph nodes: greater than or equal to 15 mm in short axis when assessed by CT scan (CT scan slice thickness must be <5 mm). The measurement should be two dimensions at axial plane. The short axis should be in perpendicular to long diameter.
6. Patient must have adequate organ function as indicated by the laboratory values. LDH less than or equal to ULN.
7. Voluntary agreement to participate as evidenced by written informed consent.
8. Female patient: agreement on contraceptive methods.
9. Male patient: agreement on contraceptive methods.
10. Life expectancy greater than or equal to 12 weeks.

Exclusion Criteria:

Patients who have not recovered to NCI CTCAE v5.0 less than or equal toGrade 1 from an adverse event (AE) due to cancer therapeutics except endocrinopathy or the chemotherapy-associated peripheral neuropathy (motor or sensory) that has recovered to CTCAE v5.0 less than or equal to Grade 2 will be allowed. The washout period for cancer therapeutic drugs should be 21 days prior to the first AI-061 dose for chemotherapy, radiation, or targeted therapy or 28 days prior to the first AI-061 administration for monoclonal antibody therapy. Best supportive care, such as thyroxine, insulin, steroid replacement treatment, blood transfusion, and therapy for non-cancer conditions are allowed.

2. Patients who are currently enrolled in any other clinical trial testing an investigational agent or device, or with concurrent other systemic cancer therapeutics.

3. Patients who are on chronic systemic steroid therapy at doses higher than 10 mg/day prednisone or equivalent within 7 days before the first treatment.

4. Patients who have active brain metastases or leptomeningeal metastases. 5. Patients who have an active infection requiring systemic IV antibiotics within 14 days prior to administration of AI-061. Regular treatment of urinary tract infection (UTI) and/or topical treatment are allowed.

6. Patients who, in the opinion of the treating Investigator, have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study or make study participation not in the best interest of the patient. The investigator should discuss this with the Sponsor.

7. Patients with known psychiatric or substance abuse disorders that in the opinion of the investigator, would interfere with cooperation with the requirements of the trial.

8. Patients who are pregnant or breastfeeding.

9. Patients with active autoimmune diseases that require immunosuppressant treatment other than 10 mg per day or lower prednisone. Patients with inflammatory bowel disease or myasthenia gravis will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 21 days after first treatment
  The number of subjects who have Dose limiting toxicity (DLT) as defined by protocol DLT criteria during the first cycle of study drug, AI-061, administration.
Maximum Toxicity Dose (MTD) | 21 day after first treatment
  Maximal tolerable dose (MTD), the study drug, AI-061, dose level that has two out of six subjects who have DLT.
Recommended Phase II Dose (RP2D) | 21 days after first treatment
  Recommended Phase II Dose (RP2D), the study drug, AI-061, dose level that is one level below MTD, or an intermediate dose level that below MTD and pre-specified in protocol. This dose level will be the RP2D.
Incidence of treatment emergent adverse events (TEAE) | From the day with first treatment to 90 days after the last treatment.
  Incidence of treatment emergent adverse events (TEAE) according to CTCAE v5.0.

SECONDARY OUTCOMES:
Cmax of AI-061 | Frequent PK samplings in cycle 1 and cycle 3, pre-dose and post-dose samples in other cycles and End of Treatment. Up to 1 year.
  The highest Serum concentration of AI-061 after IV infusion at cycle 1 and cycle 3 dosings from different timepoints after drug administration.
The serum half-life of AI-061 | Frequent PK samplings in cycle 1 and cycle 3, pre-dose and post-dose samples in other cycles and End of Treatment. Up to 1 year.
  To determine the drug concentration in serum samples that are taken in various timepoints during the treatment in order to calculate drug half life.
Objective Response Rate (ORR) | Up to 1 year.
  Objective Response Rate (ORR), evaluated by investigators on radiological images according to RECIST 1.1.
Progression free survival (PFS) | Up to 1 year.
  Progression free survival (PFS), the event is the time that diseased progressed evaluated by investigators or death occurs.
Overall survival (OS), | Up to 1 year.
  Overall survival (OS), the event is the time that all cause death occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Joshi, MD, Principal Investigator — Cancer Research South Australia
Locations (5):
- Australia (5):
  - St. Vincent's Private Hospital, Darlinghurst, New South Wales
  - Mater Misericordiae Ltd., Brisbane, Queensland
  - Tasman Oncology Research, Southport, Queensland
  - Cancer Research SA, Adelaide, South Australia
  - Southern Oncology Clinical Research Unit, Bedford Park, South Australia

IPD SHARING:
Plan to Share IPD: No